CLINICAL TRIAL: NCT00002921
Title: Evaluation of Suramin in Advanced Adrenal Cortical Carcinoma, Phase II
Brief Title: S9427, Suramin in Treating Patients With Stage III or Stage IV Adrenocortical Cancer Incurable by Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Permanently Closed Due to Lack of Accrual
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000065324; SWOG-9427 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2004-07-30 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Adrenocortical Carcinoma
Keywords: stage III adrenocortical carcinoma; stage IV adrenocortical carcinoma
MeSH Terms: conditions — Adrenocortical Carcinoma | interventions — Suramin; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Suramin (Experimental)
  Interventions: Drug: suramin; Drug: therapeutic hydrocortisone

INTERVENTIONS:
Drug: suramin
Drug: therapeutic hydrocortisone

SUMMARY:
RATIONALE: Some tumors need growth factors produced by the body to keep growing. Suramin may interfere with the growth factor and stop the tumor from growing.

PURPOSE: Phase II trial to study the effectiveness of suramin in treating patients with stage III or stage IV adrenocortical cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the response of patients with adrenocortical carcinoma treated with suramin. II. Evaluate the qualitative and quantitative toxic effects of this therapy.

OUTLINE: Patients are described according to stage, performance status, prior radiotherapy, prior surgery, and prior mitotane therapy. Patients receive suramin IV for 5 days in the first week, then twice a week for 2 weeks, and then weekly for a total of 12 weeks. Hydrocortisone is taken PO twice daily. Following a 12 week rest, patients receive a second course; those with stable or responding disease continue treatment for a maximum of four courses.

PROJECTED ACCRUAL: A maximum of 40 patients will be accrued at a rate of 6-7 per year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed adrenocortical carcinoma in Stage III or IV and incurable by surgery Bidimensionally measurable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: SWOG 0-2 Hematopoietic: WBC at least 4,000/mm3 Absolute granulocyte count at least 2,000/mm3 Platelet count at least 150,000/mm3 Prothrombin time and partial thromboplastin time no greater than upper limit of normal (ULN) Hepatic: SGOT and alkaline phosphatase no greater than 2 times ULN Renal: Creatinine clearance at least 50 mL/min Serum creatinine no greater than ULN Other: No second malignancy within 5 years except adequately treated basal cell or squamous cell carcinoma of the skin,in situ carcinoma of the cervix, or other cancer for which patient has been disease free for 5 years Not pregnant or nursing Effective contraception required of fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent biologic therapy At least 4 weeks since prior biologic therapy (one regimen only) Chemotherapy: No concurrent chemotherapy At least 4 weeks since prior mitotane No other prior chemotherapy allowed Endocrine therapy: At least 6 weeks since prior hormonal therapy No concurrent hormonal therapy Radiotherapy: At least 4 weeks since prior radiation therapy (to less than 25% of bone marrow) No concurrent radiation therapy Surgery: Prior surgery allowed in relapsed patients with no other prior treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 1997-03; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Response to suramin | From date of registration to progression or date of death from any cause, whichever came first, assessed up to four cycles

SECONDARY OUTCOMES:
Number and grade of adverse events | From date of registration until progression or date of death from any cause, whichever came first, up to four cycles

CONTACTS AND LOCATIONS:
Overall Officials: Louis E. Schroder, MD, Study Chair — Barrett Cancer Center
Locations (65):
- United States (65):
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Beckman Research Institute, City of Hope, Duarte, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Loyola University Medical Center, Maywood, Illinois
  - CCOP - Central Illinois, Springfield, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Louisiana State University Hospital - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - University of New Mexico Cancer Research & Treatment Center, Albuquerque, New Mexico
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Eastern Virginia Medical School, Norfolk, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington

REFERENCES:
- [Result] Shroder LE, Glass T, Eisenberger M, et al.: Phase II evaluation of suramin in advanced adrenal carcinoma: Southwest Oncology Group (SWOG) trial 9427. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-2361, 153b, 2001.